CLINICAL TRIAL: NCT01950962
Title: ROLE OF PHOSPHOLIPID TRANSFER PROTEINS (PLTP) ON ENDOTOXEMIA CAUSED BY BUCCAL INFLAMMATION
Acronym: TOXIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: Lafon PHRC IR 2010
Record Dates: First submitted 2013-08-27; First posted 2013-09-26 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Patients With Periodontal Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- slight periodontal disease (Other)
  Interventions: Other: Sampling of blood
- moderate periodontal disease (Other)
  Interventions: Other: Sampling of blood
- severe periodontal disease (Other)
  Interventions: Other: Sampling of blood

INTERVENTIONS:
Other: Sampling of blood

SUMMARY:
This is a transversal double-centre study. Patients will be recruited from outpatient consultations. They will have buccal inflammation caused by periodontal disease (frequent oral infections, mostly with GRAM (-) bacteria). Three groups of 80 patients, corresponding to slight, moderate and severe periodontal disease, will be formed according to the results of radiological and clinical examinations.

ELIGIBILITY:
Inclusion Criteria:

Pre-Inclusion criteria:

* Persons aged from 35 to 80 years old
* Persons who have provided written informed consent
* Patients with periodontal disease whatever the severity with at least one molar or one premolar on the dental arch
* Possibility to examine the oral cavity (patient able to open mouth)
* Possibility to do an orthopantomogram (sitting position required and patient able to clench jaws)
* Patient able to understand French
* Patient who accepts to provide fasting blood sample within the five days following the initial consultation

DEFINITIVE INCLUSION CRITERIA

- Patient present for the fasting blood sample within five days following the initial consultation Patients will be matched for sex and, as much as possible, for age in the three groups and for the severity of the periodontal disease

Exclusion Criteria:

* Persons not covered by the national health insurance agency
* Patients with a high risk of infectious endocarditis who require prophylaxis for any medical act involving blood
* Patients who have taken at least once during the 8 days preceding the definitive inclusion an anti-inflammatory dose of NSAIDS and/or a salicylate (blood sample)
* Patients who have had long-term treatment (>6 months) with corticoids at a dose of at least 15 mg per day
* Patients on antibiotics less than 15 days before the blood sample
* Patients with oral inflammation requiring treatment with antibiotics or anti-inflammatory drugs during the pre-inclusion
* Scaling during the 24 hours before the blood sample
* History of oral cancer or cancer of the pharynx
* Active cancer (patient undergoing treatment or diagnosis within the previous 5 years)
* Iatrogenic, spontaneous or therapeutic immunodepression (patient on immunosuppressants or antiretrovirals),
* Systemic or organ specific inflammatory syndrome not related to the periodontal disease

  * proven bacterial, viral or fungal Infection either developing or being treated (urinary, prostate infection)
  * Inflammatory cancer (solid tumour, malignant hemopathy)
* Pregnancy
* Impossibility to cooperate due to a psychiatric disease, dementia
* Patients unable to understand the protocol

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2014-06-12 (Actual)

PRIMARY OUTCOMES:
Score of severity of oral inflammation | up to 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France